CLINICAL TRIAL: NCT00865293
Title: Obesity and Expiratory Flow Limitation (EFL)
Brief Title: Expiratory Airflow Limitation in Subjects With Obesity
Acronym: EFL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical Center Alkmaar (Other)
Responsible Party: Dr. J.G. van den Aardweg, Medical Center Alkmaar
Other Study IDs: Obesity MCA 2009
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Obesity
Keywords: Obesity; expiratory flow limitation; EFL; posture; small airways obstruction; FOT
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obesity: Subjects with obesity, defined as BMI > 30, aged 25-60
- Control: Subjects with a BMI 18,5-25, aged 25-60

SUMMARY:
The purpose of this study is to investigate posture dependent small airway obstruction in subjects with obesity, and to study the capacity of FOT as a measurement tool for small airways obstruction.

DETAILED DESCRIPTION:
Obesity is a cause of dyspnea due to mechanical impairment of pulmonary ventilation. One of the causes of this impairment is expiratory flow limitation, which is related to decreased lung volume. As a result, obesity can cause an asthma-like symptoms. Therefore, some patients with obesity are misdiagnosed as asthma-patients, and treated with asthma medication. The effects of bronchodilators on the mechanical airway obstruction in obese subjects have not been well established.

Posture also has effect on lung volumes: they are decreased in supine position. Therefore, the interaction of obesity and supine posture might result in a larger decrease in lung volumes, and thereby a more increased airflow limitation. It has been suggested that both obesity and supine posture result in an obstruction of peripheral airways. Such an obstruction can be measured by spirometry, using the ratio of forced expiratory flow between 25 and 75% and vital capacity. This measure is highly variable, however.

The forced oscillation technique (FOT) is a non-invasive method to measure the resistance and reactant of the respiratory system. Particularly the reactance has been shown useful in the measurement of airflow limitations.

The investigators hypothesize that obesity causes a posture dependent end- expiratory airflow limitation due to a mechanical compression of lung tissue, resulting in increased resistance and reactance in the airways. Therefore, the investigators expect no protective effect of bronchodilation by salbutamol. The investigators expect that reactance measured by FOT detects differences in airflow limitation and correlates with airflow limitation as measured by spirometry.

ELIGIBILITY:
Inclusion Criteria obese population:

* Male/female, age 25-60
* BMI (body mass index) 30-40 kg/m2
* Non or ex smokers with < 10 packyears

Inclusion Criteria control population:

* Male/female, age 25-60
* BMI (body mass index) 18.5-25 kg/m2
* Non or ex smokers with <10 packyears

Exclusion Criteria obese population:

* Asthma
* COPD (FEV1/FVC<0.70)
* Reversibility >9% in FEV1 (400 microgram salbutamol)
* Other significant neuromuscular, cardiac or lung disease

Exclusion Criteria control population:

* Asthma
* COPD (FEV1/FVC<0.70)
* Other significant neuromuscular, cardiac or lung disease
* Reversibility >9% in FEV1 (400 microgram salbutamol)

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healty volunteers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-07

PRIMARY OUTCOMES:
The difference in mean values of FEF25-75/FVC between subjects with obesity and controls in supine position | 6 months

SECONDARY OUTCOMES:
The capacity of FOT as a measurement tool for small airways obstruction. The effects of posture and obesity on lung volumes, diffusion capacity, air flow limitation. The effect of bronchodilation by salbutamol on posture dependent flow limitation. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: J. G. van den Aardweg, Study Director — Medical Center Alkmaar